CLINICAL TRIAL: NCT02973516
Title: Proof of Concept Study Concerning Efficacy of P03277 MR Imaging in HCC Diagnosis, Phase IIa Clinical Study
Brief Title: Proof of Concept Study Concerning Efficacy of P03277 MR Imaging in HCC Diagnosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GDX-44-008
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Chronic Liver Disease; HepatoCellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- P03277 triphasic imaging (Experimental): P03277 will be administered in order to acquire triphasic liver imaging
  Interventions: Drug: P03277 at 0.1 mmol/kg; Drug: P03277 at 0.05 mmol/kg

INTERVENTIONS:
Drug: P03277 at 0.1 mmol/kg — P03277 will be administered at 0.1 mmol/kg BW (corresponding to 0.2 mL/kg BW) by intravenous (IV) bolus injection at 2 mL/s rate without dilution, followed by a 0.9% saline flush.
  Other Names: gadopiclenol at 0.1 mmol/kg
Drug: P03277 at 0.05 mmol/kg — P03277 will be administered at 0.05 mmol/kg BW (corresponding to 0.1 mL/kg BW) by intravenous (IV) bolus injection at 2 mL/s rate without dilution, followed by a 0.9% saline flush.
  Other Names: gadopiclenol at 0.05 mmol/kg

SUMMARY:
This study is an exploratory study aiming to collect data about diagnosis efficacy (sensitivity and specificity) of P03277 triphasic liver imaging for HCC in subjects with suspected small nodules and chronic liver disease. 30 subjects will be included, having HCC confirmed or not by previous enhanced CT and/or MRI and before any biopsy for histology analysis. The standard of reference for diagnosis will be given by the site according to their standard of care and adapted from EASL/EORTC diagnostic criteria (considering previous contrast enhanced imaging (CT and/or MRI) and/or biopsy specimen analysis given on-site and/or the more recent AFP results available). 10 additional subjects will be included to explore the diagnostic efficacy for HCC at half dose of P03277.

ELIGIBILITY:
Inclusion Criteria:

* Subject presenting with liver cirrhosis or chronic liver disease as shown by previous liver biopsy or by combination of clinical, endoscopic, biological, ultrasound parameters, and elastography
* Subject presenting with 1 to a maximum of 3 untreated hepatic nodule(s) of less than or equal to 3 cm (long axis) previously identified and/or characterized through enhanced CT and/or MRI within a maximum of 21 days before P03277 imaging, confirmed for HCC or not

Exclusion Criteria:

* Subject presenting with hepatic nodule more than 3 cm in addition to nodule(s) less than or equal to 3 cm
* Subject already treated for HCC by surgery or thermal ablation for which the resection or coagulation area is less than 2 cm from the new nodule(s)
* Subject previously treated by transarterial chemoembolization
* Subject with moderate or severe renal impairment (eGFR < 60 mL/min/1.73 m2) based on measurement done or available within the 7 days before P03277 administration and assessed after any iodinated contrast agent administration, or with dialysis end stage renal disease (ESRD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Manager, Study Director — Guerbet
Locations (2):
- France (2):
  - CHU Angers, Angers
  - Hôpital Beaujon, Clichy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 41 screened patients, one failed to meet randomization criteria and was screen failure. Therefore, 40 patients were included: 30 in Cohort 1 (0.1 mmol/kg) and 10 in Cohort 2 (0.05 mmol/kg),
Groups:
- Cohort 1: Gadopiclenol administered at 0.1 mmol/kg BW (corresponding to 0.2 mL/kg BW) by intravenous (IV) bolus injection at 2 mL/s rate without dilution, followed by a 0.9% saline flush.
- Cohort 2: Gadopiclenol administered at 0.05 mmol/kg BW (corresponding to 0.1 mL/kg BW) by intravenous (IV) bolus injection at 2 mL/s rate without dilution, followed by a 0.9% saline flush.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 30 | 10
Completed | 30 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed for the Full Analysis Set (FAS). One patient from cohort 1 was not included in the FAS for not presenting any nodule at the time of inclusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 29 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (6.5) | 60.7 (15.4) | 61 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 23 | 8 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 24 | 8 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.07 (6.08) | 27.98 (5.16) | 27.30 (5.80)

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Value Evaluation for HCC
Description: Sensitivity and specificity of diagnosis obtained by gadopiclenol imaging versus standard of reference
Time Frame: One day procedure
Population: Analysis performed on the Full Analysis Set Nodules (FASN). A total of 56 suspected nodules were characterized: 43 from cohort 1 and 13 from cohort 2.
Measure: Number; unit: percent
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 29 | 10
percent
  Sensitivity | 62 | 80
  Specificity | 86 | 100
  Accuracy | 74 | 92
  Positive predictive value | 81 | 100
  Negative predictive value | 70 | 89

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from informed consent signature up to 13 weeks after gadopiclenol administration
Description: Post-injection adverse events are reported below.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/10
Other Adverse Events (participants affected / at risk) | 8/30 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=30) | Cohort 2 (N=10)
gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=30) | Cohort 2 (N=10)
Feeling hot (General disorders) | 2 (2) | 0 (0)
Injection site coldness (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study is an exploratory study with limited number of patients included. The number of nodules in each cohort is considerably different, therefore limiting the possibility of comparison between the cohorts.

Gadopiclenol owns very high relaxivity, which prolonged the wash-out at portal or delayed phases in some cases, further clinical investigation with larger number of patients is needed to study behavior of gadopiclenol in liver imaging.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT02973516/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT02973516/SAP_001.pdf